CLINICAL TRIAL: NCT06996249
Title: Prospective Data Collection Initiative on Thoracic Malignancies - a Prospective Observational Cohort Study
Brief Title: Prospective Data Collection Initiative on Thoracic Malignancies
Acronym: DuTOC
Status: Recruiting | Type: Observational
Sponsor: Dutch Society of Physicians for Pulmonology and Tuberculosis (Other)
Responsible Party: Sponsor
Other Study IDs: Dutch Thoracic Oncology Cohort; NL-009157 / PI-01.01 (Other: CCMO)
Record Dates: First submitted 2025-05-19; First posted 2025-05-30 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer; Thoracic Cancer; Lung Cancer, Nonsmall Cell; Adenocarcinoma; Squamous Cell Carcinoma; Large Cell Lung Cancer; Thymus Cancer; Mesothelioma
Keywords: Dutch lung cancer cohort; lung cancer cohort
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma; Carcinoma, Squamous Cell; Thymus Neoplasms; Mesothelioma | interventions — Quality of Life; Tumor Burden; Histocompatibility Testing; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Biospecimen Retention: Samples With DNA — Blood and tumor tissue will be stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with a thoracic malignancy: Patients diagnosed with thoracic malignancies will be asked to participate in this cohort.
  Interventions: Behavioral: Health-related quality of life and treatment outcome questionnaires; Genetic: (Tumor) tissue and other biomaterials; Procedure: Blood samples

INTERVENTIONS:
Behavioral: Health-related quality of life and treatment outcome questionnaires — Patients who consented to the completion of questionnaires will be invited to complete questionnaires on multiple time points but not more often than once every 3 months. The length of time required for the completion of questionnaires will not exceed 150 minutes a year.
Genetic: (Tumor) tissue and other biomaterials — Tissue and other biomaterial, such as pleural effusion, is collected from material obtained during a diagnostic procedure or surgical resection. No additional interventional procedures are performed to obtain the material.
Procedure: Blood samples — Blood samples can be withdrawn on multiple time points with a maximum of 10 tubes of 10 ml per year during routine blood withdrawals (or in exceptional cases with an additional blood withdrawal).

SUMMARY:
Survival after cancer diagnosis strongly depends on local tumor extent, lymph node involvement and the presence of distant metastases. However, there remains great inter-patient variability regarding treatment outcome. A combination of molecular factors, biochemical factors, histopathological features, genomic profile, environmental factors and other clinical factors are likely to influence prognosis and treatment effect, independent from tumor stage. It is however still unclear which, how, and to what extent these factors will influence tumor recurrence and mortality in both early stage (I-III) and late stage (IV) thoracic malignancies such as lung cancer.

Although the results from prospective clinical trials will remain the backbone of evidence-based medicine, this concerns a highly selected patient population since the large majority (85%-95%) of patients with cancer do not participate in clinical trials for various reasons. It is unlikely that trial participation will significantly improve in the near future. This fact has the following implications:

1. It is highly desirable to validate the results from clinical trials in the general patient population. This is complicated by the fact that the documentation of patients treated in general practice (i.e. outside the scope of clinical trials) is largely insufficient to provide comparable patient cohorts in terms of prognostic characteristics and treatment parameters.
2. There is an ever increasing number of therapeutic interventions available for which its efficacy depends on known and unknown tumor-specific, clinical, demographic and other patient characteristics. Large numbers of patients are required to test the relevance of these variables.
3. As a result of rapid technical and drug developments, new minimally invasive treatment options such as stereotactic irradiation or ablation techniques or sublobar resections and new targeted and immunotherapeutic treatments have entered the clinic. These interventions have potentially less side effects compared to the conventional treatments. Still, these new interventions will have to prove their effectiveness, safety and superiority (or non-inferiority) in a real world setting.
4. Many hypotheses related to further optimization of personalized medicine can currently not be tested as they require a large prospective cohort of patients, and a less time-consuming and costly research infrastructure.

A prospective observational cohort study has the potential to fill the gap between prospective randomized trials (efficacy) and patients treated in general practice (effectiveness) and it will enable accrual of clinical trials (innovation).

DETAILED DESCRIPTION:
Objective:

* To start a prospective observational cohort study of patients with thoracic malignancies from their primary diagnosis until death.
* After obtaining informed consent, to prospectively collect data on medical history, comorbidities, baseline clinical parameters, imaging results, pathology results, tumor characteristics, treatment, treatment outcomes, hospital stays, interventions and (S)AEs.
* After obtaining separate informed consent for collecting data on health related quality of life and work ability, to collect data on patient reported outcome measures.
* After obtaining separate informed consent, to collect imaging, blood and (tumor) tissue material, obtained during routine practice, for observational studies or storage in the biobank.
* After obtaining separate informed consent, to collect imaging obtained during routine practice, for observational studies or AI learning.
* The cohort will serve as an infrastructure geared towards efficient, safe and comprehensive clinical evaluation of new interventions (for example multidisciplinary anti-cancer treatment, drugs or other systemic treatment, lifestyle or in follow up) for patients with thoracic malignancies when appropriate according to the Trials within Cohorts (TwiCs) design. For interventions other than standard of care a separate informed consent is mandatory.

Expected outcome:

* To provide more accurate data on the treatment and clinical outcome and patient reported outcomes of thoracic malignancies in daily practice.
* To create an infrastructure for a large variety of research purposes including but not limited to:

  * Prognostic and predictive research
  * Molecular and (epi)genetic research
  * Comparison of new therapeutic interventions for patients with thoracic malignancies, when appropriate according to the Trials within Cohorts (TwiCs) design.
  * Health care policies and cost-effectiveness studies

Study design:

A prospective observational cohort study. Patients diagnosed with thoracic malignancies will be asked to participate in this cohort. Prospectively, a limited number of variables (e.g. gender, age, histology, TNM) will in the majority of cases preferably be registered within 1-3 weeks following diagnosis. Further enrichment of the data will be done by linking this cohort to the Netherlands Cancer Registry (NCR) database (in the Netherlands clinical variables, treatment variables of all malignancies are routinely collected (Appendix I)) on a 6 monthly basis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Histo/cytopathological proof of a thoracic malignancy, or a strong suspicion (after imaging and multidisciplinary board);
* Informed consent for longitudinal observational data collection;

Exclusion Criteria:

* Mentally challenged patients that are unable to provide conscientious informed consent as determined by the investigator.
* Inability to provide a written or electronic informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with a pathological confirmed thoracic malignancy, who are recently diagnosed, or have a strong suspicion without pathological confirmation but with confirmation in the multidisciplinary tumor board in one of the participating hospitals will be asked to participate in this cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | up to 10 years

SECONDARY OUTCOMES:
Disease free survival | up to 10 years
Overall survival | up to 10 years
Health related quality of life | Baseline - 3 - 6 - 12 - 24 - 36 - ... months
  QLQc30 questionnaire with a 1 (not at all) to 4 (very much) scale
Health related quality of life | Baseline - 3 - 6 - 12 - 24 - 36 - ... months
  EQ5D questionnaire with a 1 (no problems) to 5 (not able to) scale and 0 (worst) to100 (best) measurement scale
Health related quality of life | Baseline - 3 - 6 - 12 - 24 - 36 - ... months
  LC-13 questionnaire with a 1 (not at all) to 4 (very much) scale

CONTACTS AND LOCATIONS:
Overall Officials: W.K. de Jong, Dr., Principal Investigator — UMC Utrecht
Locations (5):
- Netherlands (5):
  - Meander MC, Amersfoort
  - MUMC+, Maastricht
  - CWZ (Canisius Wilhelmina Ziekenhuis), Nijmegen
  - Erasmus MC, Rotterdam
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided
A research proposal can be submitted via DuTOC@umcutrecht.nl. A data and/or tissue requests for scientific research will be discussed and approved by a scientific committee. The scientific committee will discuss requests and the committee will subsequently decide regarding the handing out of the material and/or data.

REFERENCES:
- See also: DuTOC website — https://dutoc.nl